CLINICAL TRIAL: NCT01391572
Title: A Randomized Phase II Trial Estimating The Optimal Radiation Volume Of Postsurgical Radiation For Patients With Locoregionally Advanced Thoracic Esophageal Squamous Cell Carcinoma
Brief Title: A Trial Estimating The Optimal Radiation Volume Of Postsurgical Radiation For Patients With Esophageal Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fudan University (Other)
Collaborators: The First Affiliated Hospital of Soochow University (Other); The Affiliated Tumor Hospital of Nantong University, Nantong, Jiangsu Province, China (Other); Jiangsu Cancer Institute & Hospital (Other); Affiliated Hospital of Jiangsu University (Other); Zhejiang Cancer Hospital (Other); First Affiliated Hospital of Wenzhou Medical University (Other); Zhejiang University (Other); The First Affiliated Hospital of Anhui Medical University (Other); Anhui Provincial Hospital (Other Government); Fujian Cancer Hospital (Other Government); Shanghai Chest Hospital (Other); Shanghai Pulmonary Hospital, Shanghai, China (Other); RenJi Hospital (Other)
Responsible Party: Xiao-Long Fu / Professor, Fudan University Cancer Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2011ESO_FU_01
Record Dates: First submitted 2011-07-08; First posted 2011-07-12 (Estimated); Last update posted 2011-07-22 (Estimated); Status verified 2011-03

CONDITIONS: Esophageal Squamous Cell Carcinoma
Keywords: thoracic esophageal squamous cell carcinoma; esophagectomy; radiation; tumor bed; elective nodal irradiation
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma | interventions — Cisplatin; Fluorouracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Experimental): After esophagectomy, patients in Arm A will receive Large field radiation (tumor bed + ENI (elective nodal irradiation)) + Sequential chemotherapy
  Interventions: Radiation: enlarge irradiation volume; Drug: cisplatin; Drug: fluorouracil
- B (Active Comparator): After esophagectomy, patients in Arm B will receive small field radiation (tumor bed only) + Sequential chemotherapy
  Interventions: Radiation: Small volume radiation; Drug: cisplatin; Drug: fluorouracil

INTERVENTIONS:
Radiation: enlarge irradiation volume — In Arm A, postsurgical radiation target volume includes tumor bed and elective nodes area
  Arms: A
Radiation: Small volume radiation — In Arm B, postsurgical radiation target volume includes tumor bed only
  Arms: B
Drug: cisplatin
Drug: fluorouracil

SUMMARY:
A randomized phase II trial to estimate the optimal radiation volume of postsurgical radiation for patients with locoregionally advanced thoracic esophageal squamous cell carcinoma (T3-4, any N, M0).

DETAILED DESCRIPTION:
Patient Population:

Thoracic esophageal squamous cell carcinoma after esophagectomy with at least 15 lymph nodes removed for adequate nodal staging.

T3-4, any N, M0.

Scheme:

After esophagectomy, patients are firstly stratified by 2 factors: (1)number of lymph node metastasis (<3 or >=3) and (2)tumor resection status (R1 resection or R2 resection).

Note: Pathological R0 resection status is required for this study. So here R1 and R2 resection are not actually pathological status of resection, only clinical judgement by physician based on the chest-CT before esophagectomy.

Then patients are randomized to 2 arms:

Arm A:

Large field radiation (tumor bed + ENI (elective nodal irradiation)) + Sequential chemotherapy (4 cycles).

Arm B:

Small field radiation (tumor bed only) + Sequential chemotherapy (4 cycles).

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 and ≤70
2. Performance status 0-1
3. Weight is not less than 90% of it before operation
4. Registration within 8 weeks after esophagectomy
5. Histologically proven primary thoracic esophageal squamous cell carcinoma
6. R0 resection and number of lymph nodes dissected ≥15 after esophagectomy
7. Pathological stage of T3-4N0-3M0
8. Chest and abdominal contrast enhanced CT within 6 weeks prior to registration(PET/CT scan is selective)
9. Without supraclavicular nodes and abdominal regions nodes existed after surgery
10. Without neo-adjuvant chemotherapy and radiotherapy
11. WBC≥ 4.0X109/L ,Absolute neutrophil count (ANC) ≥ 2.0X109/L
12. Platelets ≥ 100X109/L
13. Hemoglobin ≥ 90g/L(without blood transfusion)
14. AST (SGOT)/ALT (SGPT) ≤ 2.5 x upper limit of normal, Bilirubin ≤ 1.5 x upper limit of normal
15. Creatinine ≤ 1.5 x upper limit of normal
16. Sign study-specific informed consent prior to study entry

Exclusion Criteria:

1. Multiple primary esophageal tumors
2. Prior invasive malignancy (except non-melanomatous skin cancer) unless disease free for a minimum of 2 years (For example, carcinoma in situ of the breast, oral cavity, or cervix are all permissible).
3. Severe, active comorbidity, defined as follows:

   3.1 Unstable angina and/or congestive heart failure requiring hospitalization within the last 3 months 3.2 Transmural myocardial infarction within the last 6 months 3.3 Acute bacterial or fungal infection requiring intravenous antibiotics at the time of registration 3.4 Chronic obstructive pulmonary disease exacerbation or other respiratory illness requiring hospitalization or precluding study therapy at the time of registration 3.5 Acquired immune deficiency syndrome (AIDS) based upon current CDC definition; note, however, that HIV testing is not required for entry into this protocol. The need to exclude patients with AIDS from this protocol is necessary because the treatments involved in this protocol may be significantly immunosuppressive.
4. Pregnancy or women of childbearing potential and men who are sexually active and not willing/able to use medically acceptable forms of contraception.
5. Prior systemic chemotherapy, prior radiation therapy or prior target drug therapy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2011-04; Primary Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Survival
  To evaluate if the survival outcome of postsurgical radiation with a small target volume involved tumor bed only is not worse than a large volume (tumor bed and elective nodes) for patients with locoregionally advanced thoracic esophageal squamous cell carcinoma.

SECONDARY OUTCOMES:
Safety and Tolerability
  To evaluate the incidence rate of adverse events-especially radiation-induced lung toxicity
Failure pattern
  To evaluate the rationality of radiation target volumes by analyzing the therapeutic failure patterns especially by comparing the in-field and out-of-field recurrences.

CONTACTS AND LOCATIONS:
Overall Officials: Xiao-Long Fu, M.D, Ph.D., Principal Investigator — Fudan University
Locations (1):
- Fudan University Cancer Center, Shanghai, Shanghai Municipality, China